CLINICAL TRIAL: NCT02837666
Title: Independent and Synergistic Effect of Spirulina Maxima With Exercise on General Fitness, Lipid Profile and Antioxidant Capacity in Overweight and Obese Subjects
Brief Title: Hypolipidemic and Antioxidant Capacity of Spirulina and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UACJ-ICB-2016-01
Record Dates: First submitted 2016-06-22; First posted 2016-07-19 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Dietary Supplements; WASH protein, Drosophila; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group and supplementation (Active Comparator): Supplementation with Spirulina maxima Supplementation with placebo Group with exercise program and supplementation with Spirulina maxima or placebo (4.5 g/d) in capsules during 6 weeks, then a 2 weeks washout, to finally proceed to the other treatment during 6 more weeks. During the 14 weeks of study duration every participant will have a personal isoenergetic diet.
  Interventions: Dietary Supplement: Supplementation with Spirulina maxima; Other: Washout; Other: Supplementation with placebo; Other: Isoenergetic diet; Other: Exercise program
- No exercise group and supplementation (Active Comparator): Supplementation with Spirulina maxima Supplementation with placebo Group without exercise program and supplementation with Spirulina maxima or placebo (4.5 g/d) in capsules during 6 weeks, then a 2 weeks washout, to finally proceed to the other treatment during 6 more weeks. During the 14 weeks of study duration every participant will have a personal isoenergetic diet.
  Interventions: Dietary Supplement: Supplementation with Spirulina maxima; Other: Washout; Other: Supplementation with placebo; Other: Isoenergetic diet

INTERVENTIONS:
Dietary Supplement: Supplementation with Spirulina maxima — Supplementation with Spirulina maxima (4.5 g/d) in capsules during 6 weeks.
Other: Washout — 2 weeks washout period to each study subject to avoid any possible carryover effect.
Other: Supplementation with placebo — Supplementation with placebo (4.5 g/d) in capsules during 6 weeks.
Other: Isoenergetic diet — All participants will have a personal isoenergetic diet according to their height, weight, body composition and daily physical activity during 14 weeks
Other: Exercise program — Participants are going to exercise five days a week with the following protocol: Between 5 and 10 min of heating exercise, Between 20-30 min anaerobic exercise and 20-30 min of aerobic exercise (cardiovascular exercise): walking, jogging, running and/or cycling, Three days a week aerobic intensities will be between 60% and 80% and two days between 70% and 90% of the maximum heart rate reserve, and five final minutes of stretching.
  Arms: Exercise group and supplementation

SUMMARY:
The purpose of this study is to demonstrate that Spirulina maxima intake and a dosed physical activity program will decrease, both independently and synergistically, cardiovascular risks (Dyslipidemias and oxidative stress) in overweight and obese subjects.

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of death globally, being dyslipidemias, oxidative stress, sedentary lifestyle and obesity primary risk factors. As a way to reduce cardiovascular diseases risk factors, the intake of antioxidants that come from a fruit and vegetable-rich diet or nutritional supplements, have been proposed; in this sense, the cyanobacterium Spirulina maxima is an important source of antioxidants, which is currently associated with cardiovascular protection properties. Furthermore, physical exercise at moderated intensity has protective effect exerted against cardiovascular diseases risks, mainly due to physiological adaptations, including expression of antioxidant enzymes, which stop formation and propagation of radicals, improving redox status of the organism.

There is evidence that Spirulina maxima, in addition to exercise, decreases cardiovascular diseases risks, this was mainly observed in animal models. However, no studies in humans under Spirulina maxima and exercise experimental designs proving these benefits are reported. Therefore this study will analyze the independent and synergistic effect of the intake of Spirulina maxima with a program of physical exercise at moderated intensity on general fitness, plasma lipid profile and antioxidant capacity in overweight and obese subjects.

Methods/design: Through a randomized, double blind, placebo controlled, counterbalanced crossover study design, 80 healthy overweight and obese subjects will be assessed during a 12 week isoenergetic diet, accompanied by 4.5 g/day Spirulina maxima intake and/or a systematic physical exercise program at moderate intensity. Body composition, VO2 consumption, heart rate, blood lactate, plasma concentrations of triacylglycerols, total, low and high-density lipoprotein cholesterol, antioxidant status, lipid oxidation, protein carbonyls, superoxide dismutase, catalase, glutathione, glutathione peroxidase, glutathione reductase, and paraoxonase will be assessed.

Discussion: Spirulina maxima and exercise are good alternatives to improve general fitness, to prevent or lessen dyslipidemia and oxidative stress in subjects with risk factor of chronic or noncommunicable diseases. However the independent and synergistic effect of Spirulina maxima with exercise against dyslipidemias and stress in overweight and obesity is not yet known.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (Body mass index (BMI): 25-29.9 kg/m2) and obese (BMI: > 30 kg/m2) persons

Exclusion Criteria:

* Taking drugs and/or food or vitamin supplements
* diabetes
* have a physical or electrocardiographic injury that prevents them from engaging in regular physical exercise

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Change in lipid profile | 14 weeks
  Change in plasma triacylglycerols, total cholesterol, high density lipoproteins cholesterol, and low density lipoproteins cholesterol after each treatment by using standardized enzymatic methods

SECONDARY OUTCOMES:
General fitness assessed by change in maximum oxygen consumption | 14 weeks
  Change in maximum oxygen consumption by using a gas analyzer (Cortex Metalizer 3B)
General fitness assessed by change in heart rate | 14 weeks
  Change in heart rate by using a pulsometer (Polar HT7)
General fitness assessed by change in lactate | 14 weeks
  Change in lactate concentration by using an automatized method (YSI lactate analyzer-1600)
General fitness assessed by change in body mass | 14 weeks
  Change in body fat mass and body lean mass by using pletysmography (BOD-POD)
General fitness assessed by change in blood pressure | 14 weeks
  Change in blood pressure by using an aneroid sphygmomanometer (Edimetric, Medical Technologies)
Redox status assessed by change in malondialdehyde | 14 weeks
  Change in malondialdehyde concentration by using standardized specific methods
Redox status assessed by change in protein carbonyls | 14 weeks
  Change in protein carbonyls concentration by using standardized specific methods
Redox status assessed by change in paraoxonase | 14 weeks
  Change in paraoxonase concentration by using standardized specific methods
Redox status assessed by change in superoxide dismutase | 14 weeks
  Change in superoxide dismutase concentration by using standardized specific methods
Redox status assessed by change in catalase | 14 weeks
  Change in catalase concentration by using standardized specific methods
Redox status assessed by change in glutathione | 14 weeks
  Change in glutathione concentration by using standardized specific methods
Redox status assessed by change in glutathione reductase | 14 weeks
  Change in glutathione reductase concentration by using standardized specific methods
Redox status assessed by change in glutathione peroxidase | 14 weeks
  Change in glutathione peroxidase concentration by using standardized specific methods

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Hernandez-Lepe, MS, Principal Investigator — Universidad Autonoma de Ciudad Juarez; Arnulfo Ramos-Jimenez, phD, Study Director — Universidad Autonoma de Ciudad Juarez
Locations (1):
- Universidad Autonoma de Ciudad Juarez, Juárez, Chihuahua, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Will be published in index journals
Supporting Information: Study Protocol, SAP
Time Frame: October 2019
Access Criteria: Spirulina and exercise

REFERENCES:
- [Background] Genest J, Frohlich J, Fodor G, McPherson R; Working Group on Hypercholesterolemia and Other Dyslipidemias. Recommendations for the management of dyslipidemia and the prevention of cardiovascular disease: summary of the 2003 update. CMAJ. 2003 Oct 28;169(9):921-4. No abstract available. PMID 14581310
- [Background] Ebbeling CB, Pawlak DB, Ludwig DS. Childhood obesity: public-health crisis, common sense cure. Lancet. 2002 Aug 10;360(9331):473-82. doi: 10.1016/S0140-6736(02)09678-2. PMID 12241736
- [Background] Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y, Nakayama O, Makishima M, Matsuda M, Shimomura I. Increased oxidative stress in obesity and its impact on metabolic syndrome. J Clin Invest. 2004 Dec;114(12):1752-61. doi: 10.1172/JCI21625. PMID 15599400
- [Background] Li S, Chen W, Srinivasan SR, Bond MG, Tang R, Urbina EM, Berenson GS. Childhood cardiovascular risk factors and carotid vascular changes in adulthood: the Bogalusa Heart Study. JAMA. 2003 Nov 5;290(17):2271-6. doi: 10.1001/jama.290.17.2271. PMID 14600185
- [Background] Halliwell B, Cross CE. Oxygen-derived species: their relation to human disease and environmental stress. Environ Health Perspect. 1994 Dec;102 Suppl 10(Suppl 10):5-12. doi: 10.1289/ehp.94102s105. PMID 7705305
- [Background] Schieber M, Chandel NS. ROS function in redox signaling and oxidative stress. Curr Biol. 2014 May 19;24(10):R453-62. doi: 10.1016/j.cub.2014.03.034. PMID 24845678
- [Background] Madamanchi NR, Vendrov A, Runge MS. Oxidative stress and vascular disease. Arterioscler Thromb Vasc Biol. 2005 Jan;25(1):29-38. doi: 10.1161/01.ATV.0000150649.39934.13. Epub 2004 Nov 11. PMID 15539615
- [Background] Ble-Castillo JL, Rodriguez-Hernandez A, Miranda-Zamora R, Juarez-Oropeza MA, Diaz-Zagoya JC. Arthrospira maxima prevents the acute fatty liver induced by the administration of simvastatin, ethanol and a hypercholesterolemic diet to mice. Life Sci. 2002 Apr 19;70(22):2665-73. doi: 10.1016/s0024-3205(02)01512-6. PMID 12269393
- [Background] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Background] Hosseini SM, Khosravi-Darani K, Mozafari MR. Nutritional and medical applications of spirulina microalgae. Mini Rev Med Chem. 2013 Jun 1;13(8):1231-7. doi: 10.2174/1389557511313080009. PMID 23544470
- [Background] Chamorro G, Salazar M, Favila L, Bourges H. [Pharmacology and toxicology of Spirulina alga]. Rev Invest Clin. 1996 Sep-Oct;48(5):389-99. Spanish. PMID 9005517
- [Background] Iwata K, Inayama T, Kato T. Effects of Spirulina platensis on plasma lipoprotein lipase activity in fructose-induced hyperlipidemic rats. J Nutr Sci Vitaminol (Tokyo). 1990 Apr;36(2):165-71. doi: 10.3177/jnsv.36.165. PMID 2117648
- [Background] Riss J, Decorde K, Sutra T, Delage M, Baccou JC, Jouy N, Brune JP, Oreal H, Cristol JP, Rouanet JM. Phycobiliprotein C-phycocyanin from Spirulina platensis is powerfully responsible for reducing oxidative stress and NADPH oxidase expression induced by an atherogenic diet in hamsters. J Agric Food Chem. 2007 Sep 19;55(19):7962-7. doi: 10.1021/jf070529g. Epub 2007 Aug 16. PMID 17696484
- [Background] Torres-Duran PV, Ferreira-Hermosillo A, Juarez-Oropeza MA. Antihyperlipemic and antihypertensive effects of Spirulina maxima in an open sample of Mexican population: a preliminary report. Lipids Health Dis. 2007 Nov 26;6:33. doi: 10.1186/1476-511X-6-33. PMID 18039384
- [Background] [Cholesterolemia control in Spain, 2000. A tool for cardiovascular disease prevention. Ministry of Health and Consumption, Spanish Society of Cardiology and Spanish Society of Arteriosclerosis]. Rev Esp Salud Publica. 2000 May-Jun;74(3):215-53. Spanish. PMID 10918811
- [Background] Fisher-Wellman K, Bloomer RJ. Acute exercise and oxidative stress: a 30 year history. Dyn Med. 2009 Jan 13;8:1. doi: 10.1186/1476-5918-8-1. PMID 19144121
- [Background] Morillas-Ruiz JM, Villegas Garcia JA, Lopez FJ, Vidal-Guevara ML, Zafrilla P. Effects of polyphenolic antioxidants on exercise-induced oxidative stress. Clin Nutr. 2006 Jun;25(3):444-53. doi: 10.1016/j.clnu.2005.11.007. Epub 2006 Jan 19. PMID 16426710
- [Background] Aoi W, Naito Y, Yoshikawa T. Role of oxidative stress in impaired insulin signaling associated with exercise-induced muscle damage. Free Radic Biol Med. 2013 Dec;65:1265-1272. doi: 10.1016/j.freeradbiomed.2013.09.014. Epub 2013 Sep 27. PMID 24075894
- [Background] Gomez-Cabrera MC, Domenech E, Vina J. Moderate exercise is an antioxidant: upregulation of antioxidant genes by training. Free Radic Biol Med. 2008 Jan 15;44(2):126-31. doi: 10.1016/j.freeradbiomed.2007.02.001. Epub 2007 Feb 9. PMID 18191748
- [Background] Savini I, Catani MV, Evangelista D, Gasperi V, Avigliano L. Obesity-associated oxidative stress: strategies finalized to improve redox state. Int J Mol Sci. 2013 May 21;14(5):10497-538. doi: 10.3390/ijms140510497. PMID 23698776
- [Background] Upasani CD, Khera A, Balaraman R. Effect of lead with vitamin E, C, or Spirulina on malondialdehyde, conjugated dienes and hydroperoxides in rats. Indian J Exp Biol. 2001 Jan;39(1):70-4. PMID 11349530
- [Background] Nagaoka S, Shimizu K, Kaneko H, Shibayama F, Morikawa K, Kanamaru Y, Otsuka A, Hirahashi T, Kato T. A novel protein C-phycocyanin plays a crucial role in the hypocholesterolemic action of Spirulina platensis concentrate in rats. J Nutr. 2005 Oct;135(10):2425-30. doi: 10.1093/jn/135.10.2425. PMID 16177207
- [Background] Thaakur SR, Jyothi B. Effect of spirulina maxima on the haloperidol induced tardive dyskinesia and oxidative stress in rats. J Neural Transm (Vienna). 2007 Sep;114(9):1217-25. doi: 10.1007/s00702-007-0744-2. Epub 2007 May 26. PMID 17530160
- [Background] Pescatello, Linda S., American College of Sports Medicine. Acsms Guidelines for Exercise Testing and Prescription. Wolters Kluwer/Lippincott Williams & Wilkins Health; Edición: 9th revised North American ed. 2014. 480 p
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Montoya, C. G., Ospina, C. O., Mesa, N. S., Cano, C. M., Lobo, M., Arias, P. G. G., & Pérez, B. R. Actividad antioxidante e inhibición de la peroxidación lipídica de extractos de frutos de mortiño (Vaccinium meridionale SW). Boletín Latinoamericano y del Caribe de Plantas Medicinales y Aromáticas, 2009; 8 (6): 519-528.
- [Background] Alvarez-Parrilla, E., de la Rosa, L.A., Torres-Rivas, F., Rodrigo-Garcia, J., González-Aguilar, G. Complexation of apple antioxidants: chlorogenic acid, quercetin and rutin by β-cyclodextrin (β-CD). Journal of inclusion phenomena and macrocyclic chemistry, 2005; 53 (1-2): 121-129.
- [Background] Weydert CJ, Cullen JJ. Measurement of superoxide dismutase, catalase and glutathione peroxidase in cultured cells and tissue. Nat Protoc. 2010 Jan;5(1):51-66. doi: 10.1038/nprot.2009.197. Epub 2009 Dec 17. PMID 20057381
- [Background] Jones DP, Carlson JL, Samiec PS, Sternberg P Jr, Mody VC Jr, Reed RL, Brown LA. Glutathione measurement in human plasma. Evaluation of sample collection, storage and derivatization conditions for analysis of dansyl derivatives by HPLC. Clin Chim Acta. 1998 Jul 28;275(2):175-84. doi: 10.1016/s0009-8981(98)00089-8. PMID 9721075
- [Background] Cheong SH, Kim MY, Sok DE, Hwang SY, Kim JH, Kim HR, Lee JH, Kim YB, Kim MR. Spirulina prevents atherosclerosis by reducing hypercholesterolemia in rabbits fed a high-cholesterol diet. J Nutr Sci Vitaminol (Tokyo). 2010;56(1):34-40. doi: 10.3177/jnsv.56.34. PMID 20354344
- [Background] Moura LP, Puga GM, Beck WR, Teixeira IP, Ghezzi AC, Silva GA, Mello MA. Exercise and spirulina control non-alcoholic hepatic steatosis and lipid profile in diabetic Wistar rats. Lipids Health Dis. 2011 May 15;10:77. doi: 10.1186/1476-511X-10-77. PMID 21569626
- [Background] Mazokopakis EE, Papadomanolaki MG, Fousteris AA, Kotsiris DA, Lampadakis IM, Ganotakis ES. The hepatoprotective and hypolipidemic effects of Spirulina (Arthrospira platensis) supplementation in a Cretan population with non-alcoholic fatty liver disease: a prospective pilot study. Ann Gastroenterol. 2014;27(4):387-394. PMID 25331487
- [Background] Mazokopakis EE, Starakis IK, Papadomanolaki MG, Mavroeidi NG, Ganotakis ES. The hypolipidaemic effects of Spirulina (Arthrospira platensis) supplementation in a Cretan population: a prospective study. J Sci Food Agric. 2014 Feb;94(3):432-7. doi: 10.1002/jsfa.6261. Epub 2013 Jul 10. PMID 23754631
- [Background] Anitha, L., Chandralekha, K. Effect of supplementation of spirulina on blood glucose, glycosylated hemoglobin and lipid profile of male non-insulin dependent diabetics. Asian J Exp Biol Sci; 2010; 1: 36-46.
- [Background] Ngo-Matip ME, Pieme CA, Azabji-Kenfack M, Biapa PC, Germaine N, Heike E, Moukette BM, Emmanuel K, Philippe S, Mbofung CM, Ngogang JY. Effects of Spirulina platensis supplementation on lipid profile in HIV-infected antiretroviral naive patients in Yaounde-Cameroon: a randomized trial study. Lipids Health Dis. 2014 Dec 13;13:191. doi: 10.1186/1476-511X-13-191. PMID 25496727
- [Background] Lu HK, Hsieh CC, Hsu JJ, Yang YK, Chou HN. Preventive effects of Spirulina platensis on skeletal muscle damage under exercise-induced oxidative stress. Eur J Appl Physiol. 2006 Sep;98(2):220-6. doi: 10.1007/s00421-006-0263-0. Epub 2006 Aug 30. PMID 16944194
- [Background] Kalafati M, Jamurtas AZ, Nikolaidis MG, Paschalis V, Theodorou AA, Sakellariou GK, Koutedakis Y, Kouretas D. Ergogenic and antioxidant effects of spirulina supplementation in humans. Med Sci Sports Exerc. 2010 Jan;42(1):142-51. doi: 10.1249/MSS.0b013e3181ac7a45. PMID 20010119
- [Background] Fenster CP, Weinsier RL, Darley-Usmar VM, Patel RP. Obesity, aerobic exercise, and vascular disease: the role of oxidant stress. Obes Res. 2002 Sep;10(9):964-8. doi: 10.1038/oby.2002.131. PMID 12226146
- [Background] Hernandez Lepe MA, Wall-Medrano A, Juarez-Oropeza MA, Ramos-Jimenez A, Hernandez-Torres RP. [SPIRULINA AND ITS HYPOLIPIDEMIC AND ANTIOXIDANT EFFECTS IN HUMANS: A SYSTEMATIC REVIEW]. Nutr Hosp. 2015 Aug 1;32(2):494-500. doi: 10.3305/nh.2015.32.2.9100. Spanish. PMID 26268076
- [Derived] Hernandez-Lepe MA, Olivas-Aguirre FJ, Gomez-Miranda LM, Hernandez-Torres RP, Manriquez-Torres JJ, Ramos-Jimenez A. Systematic Physical Exercise and Spirulina maxima Supplementation Improve Body Composition, Cardiorespiratory Fitness, and Blood Lipid Profile: Correlations of a Randomized Double-Blind Controlled Trial. Antioxidants (Basel). 2019 Oct 23;8(11):507. doi: 10.3390/antiox8110507. PMID 31652765
- [Derived] Hernandez-Lepe MA, Lopez-Diaz JA, Juarez-Oropeza MA, Hernandez-Torres RP, Wall-Medrano A, Ramos-Jimenez A. Effect of Arthrospira (Spirulina) maxima Supplementation and a Systematic Physical Exercise Program on the Body Composition and Cardiorespiratory Fitness of Overweight or Obese Subjects: A Double-Blind, Randomized, and Crossover Controlled Trial. Mar Drugs. 2018 Oct 1;16(10):364. doi: 10.3390/md16100364. PMID 30275428
- [Derived] Hernandez-Lepe MA, Lopez-Diaz JA, Rosa LA, Hernandez-Torres RP, Wall-Medrano A, Juarez-Oropeza MA, Pedraza-Chaverri J, Urquidez-Romero R, Ramos-Jimenez A. Double-blind randomised controlled trial of the independent and synergistic effect of Spirulina maxima with exercise (ISESE) on general fitness, lipid profile and redox status in overweight and obese subjects: study protocol. BMJ Open. 2017 Jun 23;7(6):e013744. doi: 10.1136/bmjopen-2016-013744. PMID 28645949
- See also: Statistics World Health Organization (WHO) — http://www.who.int/mediacentre/factsheets/fs317/en/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT02837666/Prot_SAP_000.pdf